CLINICAL TRIAL: NCT05291767
Title: The Effect of Moderate-Intensity Exercise on Postprandial Plasma Triglyceride Levels Following a High Fat Meal
Brief Title: High Fat Meal and Postprandial TG Levels With and Without Exercise Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel and funding issues
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Sibylle Kranz, PhD, RDN, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HSR210163
Record Dates: First submitted 2022-03-03; First posted 2022-03-23 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Ketogenic Diet; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet: high fat meal (Experimental): Participants will consume either a high fat or a high carbohydrate meal.
  Interventions: Other: Diet
- Exercise: medium intensity exercise (Experimental): After consuming the meal, participants will either exercise at moderate intensity for 30 minutes or rest.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Other: Diet — participants will consume a high fat (intervention) or high carbohydrate (control) meal.
  Other Names: High fat meal
  Arms: Diet: high fat meal
Behavioral: Exercise — participants will exercise with medium intensity under supervision for 30 minutes (intervention) or rest (control) after consuming the meal.
  Other Names: Moderate intensity exercise bout
  Arms: Exercise: medium intensity exercise

SUMMARY:
The objective of this study is to investigate whether "real-life" bouts of MIE are effective at attenuating PPTL after a meal (either a keto-type brownie (KETO) or a high carb (CON) meal of pasta and sauce), compared to non-exercise control. The primary outcome of this study is the measured change in PPTL level from baseline (fasting) to 6 hours postprandial on each activity level. We hypothesize that MIE will decrease PPTL in comparison to rest. For our secondary outcomes, we expect greater decrease in blood pressure, blood glucose, and metabolic rates after the MIE exercise bouts. Finally, we expect that KETO will be rated as more satiating.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death and disease in the United States with an overall prevalence of about 48% in adults >20 years of age. The Global Burden of Health assessment showed that CVD is largely attributed to dietary risks, followed by high systolic blood pressure (BP), high body mass index (BMI), high total cholesterol and fasting plasma triglycerides (TG), smoking, and inadequate physical activity. Increased plasma TG levels can promote atherosclerosis, atherosclerotic lesions, plaque formation, and heart attack. Consumption of high fat meals (HFM), which are very common in the American diet, likely increase postprandial triglyceride levels (PPTL), in proportion to the fat content of the meal. This is of particular concern because Americans, on average, have ~6 eating occasions throughout the day, thus maintaining a postprandial state of chronically high PPTL.

Additionally, a HFM has also been shown to negatively affect endothelial function, blood pressure, glycemic control, and resting metabolic rate. The decline in endothelial function is thought to be mediated by the oxidative stress caused by the elevated PPTL, which then contributes to proatherogenic state. Glycemic control was also found to be disrupted following consumption of a high fat meal likely due to a change in glucose absorption from the gut, glucose production in the liver, or glucose uptake from skeletal muscle. Conversely, blood pressure does not seem to be significantly affected by a high fat meal when measured up to 4 hours postprandial, although these findings are equivocal.

Recent studies have elucidated a potential role of exercise in attenuating the postprandial lipemia response via several proposed mechanisms including exercise-induced increase in fat oxidation, lipoprotein lipase (LPL) messenger ribonucleic acid (mRNA expression) and LPL activity, reduced hepatic VLDL secretions, and the creation of an energy deficit. LPL is responsible for breaking TGs down into free fatty acids, thus improving TG clearance rates. Exercise has also been shown to attenuate the increase in blood pressure and blood glucose caused by the high fat meal.

Previous studies have found that compared to a non-exercising control, moderate-intensity exercise (MIE) decreases PPTL by about 15.5% (p = 0.03) when performed prior to a HFM likely due to the increase in postprandial fat oxidation rate elicited by the exercise. Following exercise performed post-HFM, PPTL attenuation is believed to be due to a decrease in hepatic very low-density lipoprotein (VLDL) secretion, as studies have shown that hepatic VLDL concentrations decrease about 4.5 hours after exercising under post-absorptive conditions and circulating triglyceride (TG) levels of VLDL decrease by 30%. With the decrease in TG secretion, there is an increase in LPL activity that consequently increases TG clearance. Thus, as time between exercise bout and HFM consumption increases, LPL becomes an ever-increasingly important factor that further improves PPTL clearance. However, many studies have only investigated the effects of exercise prior to HFM consumption. Furthermore, many of these studies rely on exaggerated fat intake or energy expenditure in excess of the Physical Activity Guidelines for Americans. While there is one study that measured effects of exercise following a HFM, only moderate intensity (60% VO2peak) was used, and endothelial function was measured up to 4 hours postprandial the test meal and 2 hours following the exercise. However, the PPTL attenuation depends on the type of exercise, energy expenditure, intensity, energy balance, and timing relative to the HFM. Moderate intensity exercise (MIE), which is categorized as 65-75% of maximal heart rate, leads to an increase in glucose oxidation rates, which can potentially lead to a greater increase in fat oxidation in comparison to rest (no exercise) after a meal. While activity guidelines recommend engaging in either moderate or high intensity exercise, it remains unclear whether MIE changes PPTL differently after an HFM.

The objective of this study is to investigate whether "real-life" bouts of MIE are effective at attenuating PPTL after a meal (either a keto-type brownie (KETO) or a high carb (CON) meal of pasta and sauce), compared to non-exercise control. The primary outcome of this study is the measured change in PPTL level from baseline (fasting) to 6 hours postprandial on each activity level. We hypothesize that MIE will decrease PPTL in comparison to rest. For our secondary outcomes, we expect greater decrease in blood pressure, blood glucose, and metabolic rates after the MIE exercise bouts. Finally, we expect that KETO will be rated as more satiating.

This is a repeated measures cross-over design, in which all subjects will undergo rest (control) and two exercise protocols. The order of the exercise will be randomized using a traditional coin flip where each combination of flips results in a what meal/ exercise type the subject would be participating in that day. We will have an independent individual (not involved in the study) perform the study randomization and maintain the allocation schedule. Due to the nature of the exercise, blinding participants to the exercise intensity is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-45 years old

Exclusion Criteria:

* Food allergies (dairy, nuts, food dyes)
* Orthopedic or musculoskeletal contraindications to exercise
* Known cardiovascular, pulmonary, or metabolic disease
* Metal implants that may interfere with bioelectrical impedance analysis
* Answers "yes" to one or more questions on the Physical Activity Readiness Questionnaire
* Current smoker
* Blood pressure of 130/80 or higher
* Meets or exceeds American College of Sports Medicine guidelines of engaging in 150min/wk of moderate intensity exercise or 75min/wk vigorous intensity exercise Unwilling or unable to follow all aspects of the study protocol
* Female participants will have to confirm that they have a normal menstrual cycle (10-12 periods per year). If yes, they are only to participate during the follicular phase of the menstrual cycle (i.e., the week following the first day of menses).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Total Blood triglyceride levels as indicated by fasting triglycerides | Baseline
  The participant's hand will be turned upward and massaged to increase blood flow. After sanitizing, their index finger will be held in an upward position, and the lancet is placed firmly into the fingertip. The first drop of blood will be discarded. The next drop of blood, from the same fingerstick, will be placed in the device to read triglyceride levels.
Total Blood triglyceride levels as indicated by postprandial triglycerides | 2 hours postprandial
  The participant's hand will be turned upward and massaged to increase blood flow. After sanitizing, their index finger will be held in an upward position, and the lancet is placed firmly into the fingertip. The first drop of blood will be discarded. The next drop of blood, from the same fingerstick, will be placed in the device to read triglyceride levels.
Total Blood triglyceride levels as indicated by postprandial triglycerides | 4 hours postprandial
  The participant's hand will be turned upward and massaged to increase blood flow. After sanitizing, their index finger will be held in an upward position, and the lancet is placed firmly into the fingertip. The first drop of blood will be discarded. The next drop of blood, from the same fingerstick, will be placed in the device to read triglyceride levels.
Total Blood triglyceride levels as indicated by postprandial triglycerides | 5 hours postprandial
  The participant's hand will be turned upward and massaged to increase blood flow. After sanitizing, their index finger will be held in an upward position, and the lancet is placed firmly into the fingertip. The first drop of blood will be discarded. The next drop of blood, from the same fingerstick, will be placed in the device to read triglyceride levels.
Total Blood triglyceride levels as indicated by postprandial triglycerides | 6 hours postprandial
  The participant's hand will be turned upward and massaged to increase blood flow. After sanitizing, their index finger will be held in an upward position, and the lancet is placed firmly into the fingertip. The first drop of blood will be discarded. The next drop of blood, from the same fingerstick, will be placed in the device to read triglyceride levels.

SECONDARY OUTCOMES:
Blood glucose level as indicated by fasting blood glucose | Baseline
  Blood glucose will be measured using the device for finger prick blood sampling after arriving in the lab and hourly after consuming the meal.
Finger prick blood sample for blood glucose level as indicated by postprandial blood glucose | 2 hours postprandial
  Blood glucose will be measured using the device for finger prick blood sampling after arriving in the lab and hourly after consuming the meal.
Finger prick blood sample for blood glucose level as indicated by postprandial blood glucose | 4 hours postprandial
  Blood glucose will be measured using the device for finger prick blood sampling after arriving in the lab and hourly after consuming the meal.
Finger prick blood sample for blood glucose level as indicated by postprandial blood glucose | 5 hours postprandial
  Blood glucose will be measured using the device for finger prick blood sampling after arriving in the lab and hourly after consuming the meal.
Finger prick blood sample for blood glucose level as indicated by postprandial blood glucose | 6 hours postprandial
  Blood glucose will be measured using the device for finger prick blood sampling after arriving in the lab and hourly after consuming the meal.
Systolic and diastolic Blood pressure | Baseline to 6 hours postprandial in 15 minute increments
  A Bluetooth blood pressure cuff will also be given to the participant that they will wear continuously throughout the visit; data from the device will be taken at the end of the visit for 15-minute intervals.
Indirect Calorimetry: Resting Metabolic Rate | Baseline
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Resting Metabolic Rate | 2 hour postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Resting Metabolic Rate | 3 hour postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Resting Metabolic Rate | 4 hour postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Resting Metabolic Rate | 5 hour postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Resting Metabolic Rate | 6 hour postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Respiratory Exchange Ratio | Baseline
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Respiratory Exchange Ratio | 2 hours postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Respiratory Exchange Ratio | 3 hours postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Respiratory Exchange Ratio | 4 hours postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Respiratory Exchange Ratio | 5 hours postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.
Indirect Calorimetry: Respiratory Exchange Ratio | 6 hours postprandial
  Participant will lay at rest for 15 minutes prior to starting the test. A metabolic mask will then be placed over their mouth to analyze their oxygen and carbon dioxide usage to estimate their resting metabolic rate and respiratory exchange ratio. This will take about 30 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Burden of Cardiovascular Diseases Collaboration; Roth GA, Johnson CO, Abate KH, Abd-Allah F, Ahmed M, Alam K, Alam T, Alvis-Guzman N, Ansari H, Arnlov J, Atey TM, Awasthi A, Awoke T, Barac A, Barnighausen T, Bedi N, Bennett D, Bensenor I, Biadgilign S, Castaneda-Orjuela C, Catala-Lopez F, Davletov K, Dharmaratne S, Ding EL, Dubey M, Faraon EJA, Farid T, Farvid MS, Feigin V, Fernandes J, Frostad J, Gebru A, Geleijnse JM, Gona PN, Griswold M, Hailu GB, Hankey GJ, Hassen HY, Havmoeller R, Hay S, Heckbert SR, Irvine CMS, James SL, Jara D, Kasaeian A, Khan AR, Khera S, Khoja AT, Khubchandani J, Kim D, Kolte D, Lal D, Larsson A, Linn S, Lotufo PA, Magdy Abd El Razek H, Mazidi M, Meier T, Mendoza W, Mensah GA, Meretoja A, Mezgebe HB, Mirrakhimov E, Mohammed S, Moran AE, Nguyen G, Nguyen M, Ong KL, Owolabi M, Pletcher M, Pourmalek F, Purcell CA, Qorbani M, Rahman M, Rai RK, Ram U, Reitsma MB, Renzaho AMN, Rios-Blancas MJ, Safiri S, Salomon JA, Sartorius B, Sepanlou SG, Shaikh MA, Silva D, Stranges S, Tabares-Seisdedos R, Tadele Atnafu N, Thakur JS, Topor-Madry R, Truelsen T, Tuzcu EM, Tyrovolas S, Ukwaja KN, Vasankari T, Vlassov V, Vollset SE, Wakayo T, Weintraub R, Wolfe C, Workicho A, Xu G, Yadgir S, Yano Y, Yip P, Yonemoto N, Younis M, Yu C, Zaidi Z, Zaki MES, Zipkin B, Afshin A, Gakidou E, Lim SS, Mokdad AH, Naghavi M, Vos T, Murray CJL. The Burden of Cardiovascular Diseases Among US States, 1990-2016. JAMA Cardiol. 2018 May 1;3(5):375-389. doi: 10.1001/jamacardio.2018.0385. PMID 29641820
- [Background] DeSalvo KB, Olson R, Casavale KO. Dietary Guidelines for Americans. JAMA. 2016 Feb 2;315(5):457-8. doi: 10.1001/jama.2015.18396. No abstract available. PMID 26746707
- [Background] Torres N, Guevara-Cruz M, Velazquez-Villegas LA, Tovar AR. Nutrition and Atherosclerosis. Arch Med Res. 2015 Jul;46(5):408-26. doi: 10.1016/j.arcmed.2015.05.010. Epub 2015 May 29. PMID 26031780
- [Background] Patsch JR, Karlin JB, Scott LW, Smith LC, Gotto AM Jr. Inverse relationship between blood levels of high density lipoprotein subfraction 2 and magnitude of postprandial lipemia. Proc Natl Acad Sci U S A. 1983 Mar;80(5):1449-53. doi: 10.1073/pnas.80.5.1449. PMID 6402780
- [Background] Nordestgaard BG, Benn M, Schnohr P, Tybjaerg-Hansen A. Nonfasting triglycerides and risk of myocardial infarction, ischemic heart disease, and death in men and women. JAMA. 2007 Jul 18;298(3):299-308. doi: 10.1001/jama.298.3.299. PMID 17635890
- [Background] Cohn JS, McNamara JR, Cohn SD, Ordovas JM, Schaefer EJ. Postprandial plasma lipoprotein changes in human subjects of different ages. J Lipid Res. 1988 Apr;29(4):469-79. PMID 3392464
- [Background] Bae JH, Bassenge E, Kim KB, Kim YN, Kim KS, Lee HJ, Moon KC, Lee MS, Park KY, Schwemmer M. Postprandial hypertriglyceridemia impairs endothelial function by enhanced oxidant stress. Atherosclerosis. 2001 Apr;155(2):517-23. doi: 10.1016/s0021-9150(00)00601-8. PMID 11254924
- [Background] Hennig B, Toborek M, McClain CJ. High-energy diets, fatty acids and endothelial cell function: implications for atherosclerosis. J Am Coll Nutr. 2001 Apr;20(2 Suppl):97-105. doi: 10.1080/07315724.2001.10719021. PMID 11349944
- [Background] Parry SA, Smith JR, Corbett TR, Woods RM, Hulston CJ. Short-term, high-fat overfeeding impairs glycaemic control but does not alter gut hormone responses to a mixed meal tolerance test in healthy, normal-weight individuals. Br J Nutr. 2017 Jan;117(1):48-55. doi: 10.1017/S0007114516004475. Epub 2017 Jan 24. PMID 28115026
- [Background] Richter CK, Skulas-Ray AC, Gaugler TL, Lambert JD, Proctor DN, Kris-Etherton PM. Incorporating freeze-dried strawberry powder into a high-fat meal does not alter postprandial vascular function or blood markers of cardiovascular disease risk: a randomized controlled trial. Am J Clin Nutr. 2017 Feb;105(2):313-322. doi: 10.3945/ajcn.116.141804. Epub 2016 Dec 21. PMID 28003205
- [Background] Bui C, Petrofsky J, Berk L, Shavlik D, Remigio W, Montgomery S. Acute effect of a single high-fat meal on forearm blood flow, blood pressure and heart rate in healthy male Asians and Caucasians: a pilot study. Southeast Asian J Trop Med Public Health. 2010 Mar;41(2):490-500. PMID 20578534
- [Background] Heseltine D, Potter JF, Hartley G, Macdonald IA, James OF. Blood pressure, heart rate and neuroendocrine responses to a high carbohydrate and a high fat meal in healthy young subjects. Clin Sci (Lond). 1990 Nov;79(5):517-22. doi: 10.1042/cs0790517. PMID 2174321
- [Background] Jakulj F, Zernicke K, Bacon SL, van Wielingen LE, Key BL, West SG, Campbell TS. A high-fat meal increases cardiovascular reactivity to psychological stress in healthy young adults. J Nutr. 2007 Apr;137(4):935-9. doi: 10.1093/jn/137.4.935. PMID 17374657
- [Background] Freese EC, Gist NH, Cureton KJ. Effect of prior exercise on postprandial lipemia: an updated quantitative review. J Appl Physiol (1985). 2014 Jan 1;116(1):67-75. doi: 10.1152/japplphysiol.00623.2013. Epub 2013 Nov 7. PMID 24201708
- [Background] Trombold JR, Christmas KM, Machin DR, Kim IY, Coyle EF. Acute high-intensity endurance exercise is more effective than moderate-intensity exercise for attenuation of postprandial triglyceride elevation. J Appl Physiol (1985). 2013 Mar 15;114(6):792-800. doi: 10.1152/japplphysiol.01028.2012. Epub 2013 Jan 31. PMID 23372145
- [Background] Currie KD, McKelvie RS, Macdonald MJ. Flow-mediated dilation is acutely improved after high-intensity interval exercise. Med Sci Sports Exerc. 2012 Nov;44(11):2057-64. doi: 10.1249/MSS.0b013e318260ff92. PMID 22648341
- [Background] Ciolac EG, Bocchi EA, Bortolotto LA, Carvalho VO, Greve JM, Guimaraes GV. Effects of high-intensity aerobic interval training vs. moderate exercise on hemodynamic, metabolic and neuro-humoral abnormalities of young normotensive women at high familial risk for hypertension. Hypertens Res. 2010 Aug;33(8):836-43. doi: 10.1038/hr.2010.72. Epub 2010 May 7. PMID 20448634
- [Background] Batacan RB Jr, Duncan MJ, Dalbo VJ, Tucker PS, Fenning AS. Effects of high-intensity interval training on cardiometabolic health: a systematic review and meta-analysis of intervention studies. Br J Sports Med. 2017 Mar;51(6):494-503. doi: 10.1136/bjsports-2015-095841. Epub 2016 Oct 20. PMID 27797726
- [Background] Teeman CS, Kurti SP, Cull BJ, Emerson SR, Haub MD, Rosenkranz SK. Postprandial lipemic and inflammatory responses to high-fat meals: a review of the roles of acute and chronic exercise. Nutr Metab (Lond). 2016 Nov 16;13:80. doi: 10.1186/s12986-016-0142-6. eCollection 2016. PMID 27891165
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] Padilla J, Harris RA, Fly AD, Rink LD, Wallace JP. The effect of acute exercise on endothelial function following a high-fat meal. Eur J Appl Physiol. 2006 Oct;98(3):256-62. doi: 10.1007/s00421-006-0272-z. Epub 2006 Aug 3. PMID 16896723